CLINICAL TRIAL: NCT04097353
Title: Harvesting Hope for Kids: Improving Diet and Physical Activity in Childhood Cancer Survivors
Brief Title: Improving Health Behaviors for Pediatric Cancer Survivors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study recruitment of new participants was suspended during 2020 due to the Covid-19 pandemic.
Sponsor: Cynthia Gerhardt (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor-Investigator, Cynthia Gerhardt, Associate Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB1700469
Record Dates: First submitted 2019-09-10; First posted 2019-09-20 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Cancer
Keywords: Behavioral; Obesity; Neoplasm
MeSH Terms: conditions — Neoplasms; Behavior; Obesity

STUDY DESIGN:
Intervention Model Description: Families will be randomly assigned to the Harvesting Hope for Kids (HH4K) intervention or the enhanced usual care (Surviving Strong for Kids (SS4K) education group after the baseline assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Harvesting Hope for Kids (HH4K) (Experimental): Eight weekly, 60-minute sessions at a university-based farm with booster sessions. Learning is structured around fun activities to provide information about the impact of cancer treatment on children's health, as well as the importance of nutrition and physical activity in survivorship. Each session is manualized and devoted to education, a behavioral strategy applied toward a weekly goal, a cooking demonstration/taste testing, and harvesting produce from the survivor garden. Modules are offered in a group format with families together.
  Interventions: Behavioral: Harvesting Hope for Kids (HH4K)
- Surviving Strong for Kids (SS4K) (Sham Comparator): Families assigned to enhanced usual care (SS4K) group will receive education in the form of standardized guidelines for nutrition and physical activity for survivors of childhood cancer. In a one-hour session, they will learn about the impact of cancer treatment on health and the importance of nutrition and physical activity for survivors. Families will receive websites for other educational resources. They will not have access to harvesting, remote coaching, the web portal, or behavioral training to address their child's nutrition or activity.
  Interventions: Behavioral: Surviving Strong for Kids (SS4K)

INTERVENTIONS:
Behavioral: Harvesting Hope for Kids (HH4K) — Weekly meetings at university-based farm
  Arms: Harvesting Hope for Kids (HH4K)
Behavioral: Surviving Strong for Kids (SS4K) — Enhanced usual care
  Arms: Surviving Strong for Kids (SS4K)

SUMMARY:
The objective of this study is to examine the efficacy of Harvesting Hope for Kids (HH4K), a biobehavioral intervention delivered in the context of a university-based, cancer survivor garden, to increase produce intake and physical activity in survivors and caregivers.

DETAILED DESCRIPTION:
Advances in treatment have led to a rapidly growing population of over 388,500 survivors, with 13,500 new survivors expected annually. However, chronic or long-term side effects (e.g., secondary malignancies, metabolic syndrome, cardio-pulmonary toxicities) can reduce quality of life and lead to premature death. The investigators propose that diet and fitness are two critical factors for healthy survivorship given their broad impact on late effects like obesity, fatigue, and metabolic syndrome. Despite the promise of comprehensive lifestyle interventions for children who are overweight or obese, research with survivors is limited by small samples and inconsistent effects. Novel research supports a key role for the gastrointestinal (GI) microbiome in regulating weight and health outcomes, yet no studies have examined the "obesogenic" microbiome in the context of lifestyle interventions for survivors of childhood cancer. The objective of this RCT is to examine the efficacy of Harvesting Hope for Kids (HH4K), a biobehavioral intervention delivered in the context of a university-based, cancer survivor garden, to increase produce intake and physical activity in survivors and caregivers. Families will be randomized to participate in HH4K or enhanced usual care. Dietary patterns, physical activity, cardiometabolic indices, family outcomes, and GI microbiome will be assessed and the HH4K group will demonstrate greater improved than enhanced usual care.

ELIGIBILITY:
Inclusion Criteria:

* 8-12 years of age
* previously diagnosed with any type of pediatric cancer
* within 5 years post-treatment for pediatric cancer
* fluent in English, with at least 1 fluent parent
* living within 75 miles of the medical center

Exclusion Criteria:

* significant developmental disorder or cognitive difficulties that would interfere with children and caregivers completing questionnaires
* Referral to hospice or at end of life.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Fruit and Vegetable Intake | Month 0 (baseline) to Month 2 (post-intervention)
  Skin carotenoid score, with total scores ranging from 10,000-89,000+ and higher scores indicating more fruit and vegetable intake
Change in Physical Activity | Month 0 (baseline) to Month 2 (post-intervention)
  Daily step count, with higher counts indicating more physical activity

SECONDARY OUTCOMES:
Change in Child Quality of Life | Month 0 (baseline) to Month 2 (post-intervention)
  Children will complete the Pediatric Quality of Life Inventory (PedsQL), with total scores ranging from 0-92 and subscale scores ranging from 0-20/32; Higher scores indicate better quality of life
Change in Parent-rated Child Quality of Life | Month 0 (baseline) to Month 2 (post-intervention)
  Parents will complete the Pediatric Quality of Life Inventory (PedsQL) for parents, with total scores ranging from 0-92 and subscale scores ranging from 0-20/32; Higher scores indicate better quality of life
Change in Body Mass Index (BMI) | Month 0 (baseline) to Month 2 (post-intervention)
  Height, weight, and age will be combined to report BMI in kg/m^2, with lower scores indicating lower cardiometabolic risk
Change in Blood Pressure | Month 0 (baseline) to Month 2 (post-intervention)
  Lower scores indicate lower cardiometabolic risk
Change in Blood Lipids and Glucose | Month 0 (baseline) to Month 2 (post-intervention)
  Blood lipids and glucose will provide TC/HDL ratio, non-HDL cholesterol, and LDL cholesterol, with lower scores indicating lower cardiometabolic risk
Change in Microbial Diversity | Month 0 (baseline) to Month 2 (post-intervention)
  Stool samples will examine microbiome α- and β- diversity, with higher scores indicating greater microbial diversity

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Gerhardt, PhD, Principal Investigator — Abigail Wexner Research Institute at Nationwide Children's Hospital
Locations (2):
- United States (2):
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Ohio State University, Columbus, Ohio